CLINICAL TRIAL: NCT02284334
Title: Acute Effects of Dietary Glycemic Index on Lactate and Glucose Homeostasis in Individuals With Primary Mitochondrial Disease
Brief Title: Glycemic Index in Mitochondrial Disease
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 14-011156
Record Dates: First submitted 2014-10-21; First posted 2014-11-06 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Mitochondrial Diseases
Keywords: mitochondrial diseases; nutrition; glycemic index
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples obtained during MMTT.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low GI-High GI: Two study visits are separate by around one month.
  For this arm, test meal (Visit 1): low-glycemic index; test meal (Visit 2): high-glycemic index
  Interventions: Other: test meal
- High GI-Low GI: Two study visits are separate by around one month.
  For this arm, test meal (Visit 1): high-glycemic index; test meal (Visit 2): low-glycemic index
  Interventions: Other: test meal

INTERVENTIONS:
Other: test meal — low- or high-glycemic index test meal, administered during mixed meal tolerance test

SUMMARY:
The investigators are conducting a research study on nutrition in mitochondrial disease. The investigators are interested in the kind of carbohydrates that people eat. Carbohydrates are an important source of energy. Certain kinds of carbohydrates tend to raise blood sugar more in healthy people, and others tend to raise blood sugar less in healthy people. The investigators would like to know if by eating the "right" type of carbohydrate, people with mitochondrial disease can avoid high lactate levels, high blood sugar levels, and, later, low blood sugars.

In this study, this question will be answered by finding out how people with mitochondrial disease respond to two different test meals containing different kinds of carbohydrates. Neither participants nor the investigators will know which kind of test meal participants are eating.

DETAILED DESCRIPTION:
This research study involves two study visits at CHOP, each around 6 to 8 hours long. The time the visit takes can depend on how long it takes to complete the study procedures listed. This can be different from person to person. The length of time between Visit #1 and Visit #2 will be between 2 weeks and 3 months. Overall study participation will not exceed 6 months.

The study involves the following tests and procedures. These happen at each of the two visits:

* Interviews: A team member will take the participant's medical history, along with a listing of any medications s/he is taking. Throughout the study the participant will be asked to report if s/he thinks that anything bad has happened as a result of the study.
* 3-day diet record: The investigator will collect the record the participant made of everything s/he ate for the 3 days before the study visit.
* Physical Examination: The investigators will measure the participant's weight, height, blood pressure, heart rate and respiratory rate, and waist circumference. If the participant is under age 21 years, a pediatric endocrinologist will check how far s/he is along in puberty. For both boys and girls, pubic hair growth will be checked. For girls, breast development will be checked. For boys, testicular development will be checked. This examination will take approximately 2 minutes and will be done in a private room.
* Pregnancy Test (female subjects): If a female participant is eleven years old or older and/or has already started having periods, she will be asked to take a pregnancy test before starting this study.
* Questionnaires: Investigators will ask the participant to fill out questionnaires on his/her physical function and well-being. These are designed for people with mitochondrial disease (or for parents of children with mitochondrial disease). They should take around 20 minutes.
* Pre-Test Fast: The participant will not be able to eat or drink anything except plain, unflavored water (i.e., you will "fast") for at least 4 hours before the mixed-meal tolerance test starts. S/he will get the test meal at that time. S/he will receive a recommendation when the visit is scheduled when to begin fasting. This recommendation is designed for no more than 10 hours of fasting, or the participant's longest usual overnight fast, whichever is shorter.
* Mixed Meal Tolerance Test (MMTT): The test includes placement of an intravenous (IV) line in the participant's arm/hand to make taking the blood samples easier. With the IV in place, the participant will not need to be stuck again for any further blood draws, unless the IV stops working. If s/he prefers, a numbing cream can be placed on your skin for about 45 minutes before this test to numb the area. Once the IV is in place, the participant will receive a test "shake". S/he will have about 30 minutes to finish the shake. Over the next 4 hours, blood will be drawn every 30 minutes from the IV line. The total amount of blood drawn for the MMTT will be a little less than 2 tablespoons.
* Cognitive Testing: Two times during the MMTT participants will be asked to perform some testing on a computer (for example, pressing a button as soon as you see a symbol appear). Each test will take around 14 minutes and tests things like attention and reaction time. We will show you how these tests work before the MMTT.
* Dual Energy X-ray Absorptiometry (DXA) Scan: A special x-ray of the body called a DXA scan will be done to measure the amount of fat and lean (non-fat) tissue in the participant's body. During the DXA scan, the participant will be asked to lie flat on your back on a table as the scanning machine moves above the participant's body. The DXA scan is like an X-ray, and takes about 5-10 minutes. This test is painless and does not involve any needles.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 15 kg
* Girls ≥ 11 years of age and/or who have achieved menarche must have a negative urine pregnancy test.
* Genetic and/or biochemical diagnosis of mitochondrial disease.
* Eat meals by mouth during the day.

Exclusion Criteria:

* Diabetes requiring insulin.
* Receive daytime total parenteral nutrition (TPN) and/or continuous enteral feedings.
* Prescribed dietary contraindication to mixed meal tolerance testing, e.g., ketogenic diet.
* Any investigational drug use within 30 days prior to enrollment.
* Pregnant or lactating females.
* Persons unable to fast for at least 4 hours.
* Persons who may be allergic to the test meals (shakes).
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-adherent to study schedules or procedures.

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with mitochondrial diseases, from existing observational cohort study and/or CHOP Genetics/Metabolism clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
lactate area under the curve (AUC) for 3 hours after MMTT | visit 1 (baseline, 0 months), visit 2 (around 1 month)
  within-subject change in lactate area under the curve (AUC) for 3 hours (low- vs. high- glycemic index)

SECONDARY OUTCOMES:
hypoglycemia (< 70 mg/dL) post-MMTT | visit 1 (baseline, 0 months), visit 2 (around 1 month)
glucose area under the curve (AUC) for 3 hours after MMTT | visit 1 (baseline, 0 months), visit 2 (around 1 month)
  within-subject change in glucose area under the curve (AUC) for 3 hours (low- vs. high- glycemic index)
insulin area under the curve (AUC) for 3 hours after MMTT | visit 1 (baseline, 0 months), visit 2 (around 1 month)
  within-subject change in insulin area under the curve (AUC) for 3 hours (low- vs. high- glycemic index)
combined index of attention (CPT-III) during MMTT | visit 1 (baseline, 0 months), visit 2 (around 1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States